CLINICAL TRIAL: NCT03868787
Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Control During Cervical Dilator Placement Prior to Dilation and Evacuation: A Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Control During Cervical Dilator Placement Prior to Dilation and Evacuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ashley Turner, MD (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor-Investigator, Ashley Turner, MD, Co-investigator, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00209157
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: The experimental group will have an active TENS unit - Chattanooga Primera - and the control group will have a sham TENS unit. The sham TENS will be the same unit without the true TENS electrical connections. The true TENS unit consists of the active unit and electrode pads connected to the unit via direct wires. The sham group will be given the active unit and have electrode pads placed but without wire connections. These participants will be told the device is a wireless device. They will also be told they may or may not feel sensation from the TENS. This will allow the device to be powered on and run in the same manner as the active group, but will not allow for electrical transmission between the unit and electrodes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS (Experimental): The active TENS unit consists of the active unit and electrode pads connected to the unit via direct wires. The program that will be used is a high frequency (80Hz) program that runs for an hour in duration. It will be initiated 5 minutes prior to speculum placement. Participants will be instructed to increase the amplitude of the current as needed to provide analgesia but avoiding discomfort from the TENS stimulation
  Interventions: Device: TENS
- Sham TENS (Sham Comparator): The sham TENS will be the same unit without the true TENS electrical connections. The sham group will be given the active unit and have electrode pads placed but without wire connections. These participants will be told the device is a wireless device. They will also be told they may or may not feel sensation from the TENS. This will allow the device to be powered on and run in the same manner as the active group, but will not allow for electrical transmission between the unit and electrodes
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: TENS — TENS units are small, inexpensive, portable, battery-powered devices which deliver mild, alternating electrical currents via electrodes positioned on the skin near the anticipated dermatomal distribution of pain.
  Arms: Active TENS
Device: Sham TENS — Non-active TENS unit
  Arms: Sham TENS

SUMMARY:
This study evaluates the use of Transcutaneous Electrical Nerve Stimulation (TENS) as a method of pain control during osmotic dilator insertion prior to dilation and evacuation. Half the group will have an active TENS unit and half will have a sham or placebo TENS unit.

DETAILED DESCRIPTION:
Dilation and Evacuation is the most common method of second trimester abortion. Studies have shown that adequate cervical preparation is necessary for the procedure to be performed safely and reduce the risk of complications. However, in the majority of cases the placement of these dilators is done with minimal pain management options.

Transcutaneous electrical nerve stimulation (TENS) has been used in pain relief since 1965, when Melzack and Walls proposed using electrical stimulation as analgesia based on the gate control theory of pain relief. TENS units are small, inexpensive, portable, battery-powered devices which deliver mild, alternating electrical currents via electrodes positioned on the skin near the anticipated dermatomal distribution of pain. The parameters of pulse frequency and pulse intensity are adjustable and linked to TENS efficacy. They overall have a favorable safety profile. Contraindications include electronic implants, such as cardiac pacemakers and implantable cardioverter defibrillators.

Two main theories have been proposed regarding how TENS provides analgesia. According to the "gate control" theory, neuromodulation may activate large myelinated afferent nerve fibers in the dorsal horn to inhibit transmission in primary afferent nociceptive fibers. The inhibitory input from the large myelinated afferent fibers is thought to be able to "close the gate" to prevent transmission of pain sensation. The endorphin-mediated theory of pain relief states that a stimulus outside the central nervous system can raise the level of endogenous endorphins and therefore provide analgesia.

The proposed study is a single-blinded randomized controlled trial studying use of TENS for pain control during initial dilator insertion prior to dilation and evacuation. The participants will be randomized in a 1:1 randomization scheme using opaque, sequentially numbered envelopes following consent. The experimental group will have an active TENS unit - Chattanooga Primera - and the control group will have a sham TENS unit. The sham TENS will be the same unit without the true TENS electrical connections. The true TENS unit consists of the active unit and electrode pads connected to the unit via direct wires. The sham group will be given the active unit and have electrode pads placed but without wire connections. These participants will be told the device is a wireless device. They will also be told they may or may not feel sensation from the TENS. This will allow the device to be powered on and run in the same manner as the active group, but will not allow for electrical transmission between the unit and electrodes.

Based on power calculations, 56 participants are needed to detect a 20mm difference in VAS score with a standard deviation of 30mm. This is based on both minimum clinically significant difference in pain scores as well as previous studies regarding pain during dilator insertion. We will attempt to recruit 70 patients to account for possible TENS unit misuse or study dropout.

Eligible patients will have two electrodes will be placed in the suprapubic area in the bilateral lower quadrants. The program that will be used is a high frequency (80Hz) program that runs for an hour in duration. It will be initiated 5 minutes prior to speculum placement. Participants will be instructed to increase the amplitude of the current as needed to provide analgesia but avoiding discomfort from the TENS stimulation. All participants will receive a paracervical block of 20mL 1% lidocaine with sodium bicarbonate followed by rigid dilation and dilator placement per standard cervical preparation protocol. Participants will complete 100mm VAS immediately following dilator placement. VAS is a 100mm line on sheet of paper with 0 being no pain and 100mm being worst pain of their life. The number of dilators, type of dilators, and use of adjunctive mifepristone/misoprostol will be according to providers' clinical judgement. Dilator placement will be performed by either Family Planning Fellow, PGY-3 OB/GYN resident, or Nurse Practitioner. All participants will receive prescriptions for twenty tablets of ibuprofen (600mg) and twelve tablets of hydrocodone/acetaminophen 5/325, which is the standard post-dilator insertion pain protocol for this clinic site. Participants will be allowed to leave prior to the end of the initial one-hour program. They will be sent home with instructions of how to run the TENS unit as needed for pain control.

Following the initial hour of use patients can re-activate the TENS unit as often as desired, using the same program. Participants will be given a log to record when TENS unit was used and whether additional pain medications were taken. They will return their completed log and bring pill bottles on the day of surgery to confirm medications used.

Of note, in our practice a second set of cervical dilators is often placed 6 hours after first set in patients over 20 weeks gestation. During this placement the first set is removed, further rigid dilation is performed, and new dilators are placed per standard cervical preparation protocol. Pain score on 100mm VAS will be recorded following this dilator placement as well as a secondary outcome. Participants will run the TENS unit in the same manner as the initial dilator placement for dilator exchange.

On the day of surgery participants will record their highest interval pain score on 100mm VAS. They will also be asked their satisfaction with the TENS device. The TENS unit will be returned on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years of age
2. Gestational age between 14 weeks and 23 weeks 6 days
3. Willing and able to sign an informed consent in English
4. No contraindications to TENS

Exclusion Criteria:

1. Incarceration
2. Preterm Premature Rupture of Membranes or evidence of intra-amniotic infection
3. Presence of implanted cardiac device
4. Lack of sensation to touch on area of electrode placement
5. Prior TENS use
6. Opioid dependence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne McCloskey, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Center for Family Planning and Contraception, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binder P, Gustafsson A, Uvnas-Moberg K, Nissen E. Hi-TENS combined with PCA-morphine as post caesarean pain relief. Midwifery. 2011 Aug;27(4):547-52. doi: 10.1016/j.midw.2010.05.002. Epub 2010 Jul 7. PMID 20615594
- [Background] De Angelis C, Perrone G, Santoro G, Nofroni I, Zichella L. Suppression of pelvic pain during hysteroscopy with a transcutaneous electrical nerve stimulation device. Fertil Steril. 2003 Jun;79(6):1422-7. doi: 10.1016/s0015-0282(03)00363-7. PMID 12798892
- [Background] ELECTROPHYSICAL AGENTS - Contraindications And Precautions: An Evidence-Based Approach To Clinical Decision Making In Physical Therapy. Physiother Can. 2010 Fall;62(5):1-80. doi: 10.3138/ptc.62.5. Epub 2011 Jan 5. No abstract available. PMID 21886384
- [Background] Olsen MF, Elden H, Janson ED, Lilja H, Stener-Victorin E. A comparison of high- versus low-intensity, high-frequency transcutaneous electric nerve stimulation for painful postpartum uterine contractions. Acta Obstet Gynecol Scand. 2007;86(3):310-4. doi: 10.1080/00016340601040928. PMID 17364305
- [Background] Johnson MI, Paley CA, Howe TE, Sluka KA. Transcutaneous electrical nerve stimulation for acute pain. Cochrane Database Syst Rev. 2015 Jun 15;2015(6):CD006142. doi: 10.1002/14651858.CD006142.pub3. PMID 26075732
- [Background] Kayman-Kose S, Arioz DT, Toktas H, Koken G, Kanat-Pektas M, Kose M, Yilmazer M. Transcutaneous electrical nerve stimulation (TENS) for pain control after vaginal delivery and cesarean section. J Matern Fetal Neonatal Med. 2014 Oct;27(15):1572-5. doi: 10.3109/14767058.2013.870549. Epub 2014 Jan 8. PMID 24283391
- [Background] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724
- [Background] Platon B, Andrell P, Raner C, Rudolph M, Dvoretsky A, Mannheimer C. High-frequency, high-intensity transcutaneous electrical nerve stimulation as treatment of pain after surgical abortion. Pain. 2010 Jan;148(1):114-119. doi: 10.1016/j.pain.2009.10.023. Epub 2009 Dec 2. PMID 19959293
- [Background] Proctor ML, Smith CA, Farquhar CM, Stones RW. Transcutaneous electrical nerve stimulation and acupuncture for primary dysmenorrhoea. Cochrane Database Syst Rev. 2002;2002(1):CD002123. doi: 10.1002/14651858.CD002123. PMID 11869624
- [Background] Soon R, Tschann M, Salcedo J, Stevens K, Ahn HJ, Kaneshiro B. Paracervical Block for Laminaria Insertion Before Second-Trimester Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2017 Aug;130(2):387-392. doi: 10.1097/AOG.0000000000002149. PMID 28697113
- [Background] de Sousa L, Gomes-Sponholz FA, Nakano AM. Transcutaneous electrical nerve stimulation for the relief of post-partum uterine contraction pain during breast-feeding: a randomized clinical trial. J Obstet Gynaecol Res. 2014 May;40(5):1317-23. doi: 10.1111/jog.12345. Epub 2014 Apr 21. PMID 24750301
- [Background] Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014 May;4(3):197-209. doi: 10.2217/pmt.14.13. PMID 24953072

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active TENS | Sham TENS
Started | 37 | 37
Completed | 35 | 36
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: 37 participants began study in each arm. Two withdrew from the active group and one from the sham group due to not wanting to participate in the study further
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TENS | Sham TENS | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Median (Full Range); unit: years] | 32 [20 to 40] | 34 [19 to 44] | 33 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 26 | 23 | 49
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74
Parity [Median (Full Range); unit: Living Children] | 1 [0 to 4] | 1 [0 to 4] | 1 [0 to 4]
BMI [Median (Full Range); unit: Kg/m^2] | 26.7 [16.9 to 53.5] | 25.5 [18.5 to 42.2] | 25.7 [16.9 to 53.5]

OUTCOME MEASURES:

1. Primary Outcome: Pain Following Dilator Placement
Description: Self-reported pain on 100mm visual analog scale (VAS) immediately following dilator placement. Range is from 0mm to 100mm, with 0mm being the least amount of pain (minimum score) and 100mm being the greatest (maximum score). Higher values are considered a worse outcome.
Time Frame: within 5 mins after dilator placement procedure
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 35 | 36
units on a scale | 64 [7 to 94] | 60.5 [6 to 100]

2. Secondary Outcome: Interval Pain
Description: Self-reported highest level of pain between dilator placement and D&E on 100mm visual analog scale (VAS). Range is from 0mm to 100mm, with 0mm being the least amount of pain (minimum score) and 100mm being the greatest (maximum score). Higher values are considered a worse outcome.
Time Frame: 5 mins after dilator placement to 36 hours after dilator placement
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 35 | 36
units on a scale | 39 [0 to 89] | 55 [0 to 100]

3. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with device based on 4 questions with 5 point Likert scale. Minimum value is 1, maximum is 5. Higher score is a better outcome.
Time Frame: 24-36 hours after dilator placement, immediately prior to D&E
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Active TENS | Sham TENS
Number analyzed (Participants) | 35 | 36
score on a scale
  Pain control | 4 [2 to 5] | 3 [1 to 5]
  Comfort | 5 [1 to 5] | 4 [1 to 5]
  Ease of use | 2 [1 to 5] | 4 [1 to 5]
  Would you use again | 3 [1 to 5] | 2 [1 to 5]

ADVERSE EVENTS:
Time Frame: Data was collected from the 24 hours during which patients were using the TENS device
Description: No adverse events
Arm/Group | Active TENS | Sham TENS
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

LIMITATIONS AND CAVEATS:
Small study Population mostly white, non-hispanic Mostly terminating for fetal anomaly, which does not make up the vast majority of terminations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT03868787/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT03868787/ICF_002.pdf